CLINICAL TRIAL: NCT01875406
Title: Diagnosis of Sacroiliac Joint Pain: Predictive Value of a Diagnostic SIJ Injection Following a Composite of 3 Diagnostic Tests and a Pain Referral Diagram
Brief Title: a Diagnostic SIJ Injection Following a Composite of 3 Diagnostic Tests and a Pain Referral Diagram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-416
Record Dates: First submitted 2013-06-05; First posted 2013-06-11 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Sacroiliac Injection
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diagnostic exercises (Experimental): The three diagnostic exercises will be administered in random order to minimize effects of order and period on the results. Enrollment logs and study randomization will be administered electronically via a respective REDCap data modules. The enrollment, randomization and diagnostic tests will be administered by research coordinator or PI. The patients will be independently evaluated and scheduled for SIJ injection by Cleveland Clinic pain clinic staff and fellow pain physicians.
  Interventions: Other: diagnostic exercises

INTERVENTIONS:
Other: diagnostic exercises
  Other Names: questionnaires; pain surveys

SUMMARY:
The purpose of this study is to determine the predictive value of a composite of 3 simple clinically practical diagnostic tests (Mekhail's test, Patrick's and Thigh thrust) combined with a pain referral diagram in predicting response to a single diagnostic SIJ injection.

DETAILED DESCRIPTION:
The purpose of this study is to determine the predictive value of a composite of 3 simple, clinically practical, diagnostic tests (Mekhail, Patrick's and Thigh thrust) combined with a pain referral diagram in predicting response to a single diagnostic SIJ injection. The goal is to test these 3 tests and compare their predictive value to the 6 tests commonly reported in the literature in order to provide a clinician with clinically practical special tests to aide in the diagnosis and treatment of SIJ mediated pain. . Specifically, we seek to evaluate the prognostic capacity for a series of three clinical tests (Mekhail's Test, thigh thrust and Patrick's Test) combined with a pain referral diagram to accurately predict the response (change in VAS) of a single diagnostic Sacroiliac joint and extra-capsular joint injection.

ELIGIBILITY:
Inclusion Criteria:

* any patient presenting with low back pain with or without radicular symptoms, regardless of prior history of back surgery from 18-90 years old whom after being evaluated by an independent clinician in the Cleveland Clinic pain clinic has been scheduled for a diagnostic SIJ injection.

Exclusion Criteria:

* any patient less than 18 or greater than 90 years old, has any medical condition that would not allow them to complete the study, diagnosis of any recent fractures in the lumbar spine, recent infection, pregnancy, taking anticoagulants.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
validity of assessments | Day 1
  The goal is to test these 3 tests and compare their predictive value to the 6 tests commonly reported in the literature in order to provide a clinician with clinically practical special tests to aide in the diagnosis and treatment of Sacroiliac joint (SIJ) mediated pain.

SECONDARY OUTCOMES:
prognostic assessment | Day 1
  Specifically, we seek to evaluate the prognostic capacity for a series of three clinical tests (Mekhail's Test, thigh thrust and Patrick's Test) combined with a pain referral diagram to accurately predict the response of a single diagnostic Sacroiliac joint and extra-capsular joint injection.

CONTACTS AND LOCATIONS:
Overall Officials: Maged Guirguis, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No